CLINICAL TRIAL: NCT07232433
Title: Safety and Efficacy Evaluation of Cryoablation for Ground-Glass Nodules: A Single-Arm, Prospective, Open-Label Clinical Study
Brief Title: Safety and Efficacy Evaluation of Cryoablation in the Treatment of Ground-Glass Nodules
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Hecheng Li M.D., Ph.D, Chair of Department of Thoracic Surgery, Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RTS-027
Record Dates: First submitted 2025-09-27; First posted 2025-11-18 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Cryosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cryoablation group (Experimental)
  Interventions: Procedure: Cryoablation

INTERVENTIONS:
Procedure: Cryoablation — Following enrollment, patients will undergo comprehensive preoperative evaluations, including thoracic computed tomography (CT), echocardiography, pulmonary function tests, electrocardiography, and laboratory blood tests, to confirm eligibility and exclude any contraindications. Eligible patients will be admitted for cryoablation, performed either percutaneously or under electromagnetic navigation bronchoscopy (ENB) guidance, followed by a structured postoperative follow-up regimen.

SUMMARY:
Lung cancer is the leading cause of cancer-related mortality worldwide, making early diagnosis and intervention critical. With the widespread adoption of low-dose computed tomography (LDCT) screening, the detection rate of pulmonary ground-glass nodules (GGNs) has increased significantly. Although video-assisted thoracoscopic surgery (VATS) remains the standard treatment for early-stage lung cancer, a considerable proportion of patients are ineligible for surgery due to advanced age, impaired cardiopulmonary function, or multiple nodules. Cryoablation, a minimally invasive ablation technique, uses ultra-low temperatures to induce tumor cell death. It offers distinct advantages, including well-defined ablation margins, reduced procedural pain, preservation of adjacent healthy structures, and potential immune activation, providing an important alternative for this patient population. However, the safety and long-term efficacy of cryoablation for GGNs require further high-quality clinical evidence.

This study aims to conduct a prospective, single-center, open-label clinical trial to systematically evaluate the feasibility and outcomes of cryoablation (percutaneous or electromagnetic navigation bronchoscopy [ENB]-guided) for treating pulmonary GGNs. We plan to enroll 90 patients who meet the following criteria: pathologically or multidisciplinary team (MDT)-confirmed malignancy, GGN size ranging from 6-30 mm, solid component ratio <25%, unsuitability for or refusal of surgery/radiotherapy, and an Eastern Cooperative Oncology Group (ECOG) performance status of 0-1. The primary endpoint is the 2-year local recurrence rate after ablation. Secondary endpoints include the 5-year local recurrence rate, 3- and 5-year disease-free survival (DFS) rates, technical success rate (ablation completion), perioperative complications (e.g., pneumothorax, hemorrhage, infection), postoperative pulmonary function, pain scores, length of hospital stay, and treatment-related costs. The results of this study will provide critical clinical evidence to support the use of cryoablation for GGNs, optimize patient selection criteria, and promote the advancement of this minimally invasive technique.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Malignancy confirmed by histopathology or multidisciplinary team (MDT) discussion.

For a solitary GGN: size between 6-30 mm. For multiple GGNs: each measuring 6-30 mm, with no more than 3 nodules deemed to require treatment upon MDT consensus.

* Patient is ineligible for or unwilling to undergo video-assisted thoracoscopic surgery (VATS).
* Patient is ineligible for or declines radiotherapy or stereotactic body radiotherapy (SBRT).
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* The subject demonstrates good compliance and has voluntarily provided written informed consent to participate.

Exclusion Criteria:

* Presence of severe cardiac, pulmonary, hepatic, or renal dysfunction, rendering the patient ineligible for general anesthesia.
* Contraindication to either bronchoscopy or computed tomography (CT)-guided percutaneous puncture.
* High risk associated with percutaneous puncture for at least one target lesion, or absence of a feasible access route as determined by pre-procedural bronchoscopic path planning.
* Platelet count < 50 × 10⁹/L, or presence of an uncorrectable bleeding diathesis or coagulation disorder (prothrombin time > 18 seconds, or prothrombin activity < 40%).
* Concurrent participation in another interventional clinical trial, or anticipation of requiring additional antitumor therapy outside the scope of this study during the trial period.
* Any other condition deemed by the investigator to render the patient unsuitable for study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-11-21 (Actual); Primary Completion 2028-10-01 (Estimated); Study Completion 2030-10 (Estimated)

PRIMARY OUTCOMES:
2-Year Local Recurrence Rate | At 2 Years Post-Treatment

SECONDARY OUTCOMES:
Technical Success Rate | Perioperative

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Deidentified participant data
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: With publication
Access Criteria: Interested investigators will be required to submit a formal letter of intent outlining research aims, rationale, and approach. Furthermore, documentation of local IRB approval, including a description of type of review, should be submitted with the data request.